CLINICAL TRIAL: NCT01743885
Title: Efficacy and Safety of Propranolol Versus Acebutolol on the Proliferative Phase of Infantile Hemangioma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8638
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Hemangioma
Keywords: Hemangioma; Beta-blocker; Acebutolol; Propranolol; Randomized controlled trial; Infants
MeSH Terms: conditions — Hemangioma | interventions — Acebutolol; Propranolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- propanolol (Active Comparator): Propanolol (Syprol:oral solution)
  Interventions: Drug: Propanolol
- Acebutolol (Active Comparator): Acebutolol (Sectral:oral solution)
  Interventions: Drug: Acebutolol

INTERVENTIONS:
Drug: Acebutolol — 10 mg/kg/jour in 2 doses during 90 days after gradual increase of doses in the first week
  Other Names: Sectral
  Arms: Acebutolol
Drug: Propanolol — 3 mg/kg/jour in 3 doses during 90 days after gradual increase of doses in the first week
  Other Names: Syprol
  Arms: propanolol

SUMMARY:
There is no effective treatment for hemangioma regardless of immediate severity. That is in this respect a orphan disease. These hemangiomas, sometimes large, will have a phase of proliferation of several months (very scary for parents) and regression over several years. The natural history is peppered with local complications (ulcers) and aesthetic and psychological sequelae (sometimes major for the child and the family). The effects of acebutolol and propranolol on the proliferative hemangiomas were discovered accidentally by two French teams (Montpellier for acebutolol and Bordeaux for propranolol). Acebutolol and propranolol have been used for many years for the treatment of hypertension and congenital heart disease, including infants, with few side effects. The effects of acebutolol and propranolol were immediately visible with reduced volume and skin whitening of the hemangioma. In a preliminary study, acebutolol was administered to 20 patients in Montpellier with big regression of hemangiomas. The aim of the study was to compare the clinical efficacy of acebutolol (10mg/Kg/jour) and propranolol (3mg/Kg/j) on the proliferative phase of infantile hemangioma in infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 6 months
* Presenting a hemangioma with the following characteristics:

  * subcutaneous and / or cutaneous
  * minimum diameter of 1.5cm on face, 5cm outside face and 3cm if it is ulcerated.
  * without functional impairment requiring treatment or vital corticosteroid
* Consent of both parents (or the person having parental authority in families)
* Which at least one parent is a beneficiary of a social security system.

Exclusion Criteria:

* Indication of treatment with corticosteroids for an indication other than hemangioma
* Indication of treatment with beta-blocker for another indication that the hemangioma
* Infant presenting cons-indications for the administration of acebutolol or propranolol:

  * Asthma and chronic obstructive pulmonary disease in their severe forms.
  * Heart failure controlled by treatment.
  * Cardiogenic shock
  * Prinzmetal Angina
  * Bradycardia (<80 beats / min at rest the first month <70/minute from 1 to 6 month).
  * Raynaud's phenomenon and peripheral arterial disorders in their severe forms.
  * Pheochromocytoma untreated.
  * Low blood pressure (blood pressure <60/30 mmHg before 6 months)
  * Hypersensitivity to acebutolol or propranolol
  * History of anaphylactic reaction.
  * Treatment with amiodarone and / or calcium channel blockers.
  * Congenital heart disease outside inter auricular communication (CIA) or inter ventricular communication (CIV) insignificant

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hemangioma size | 3 months
  It will be evaluated using a VAS (visual analogue scale) on a series of photos at Day 0, Day 30 and Day 90

SECONDARY OUTCOMES:
Tolerance of treatment | 3 months
  All adverse events are collected at each visited
Proportion of patients requiring treatment with corticosteroids because of the evolution of a 'serious' hemangioma | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Bigorre, PH, Principal Investigator — UH Montpellier
Locations (4):
- France (4):
  - UH Lyon, Lyon
  - UH Marseill, Marseille
  - Chirurgy Plastic Department, Montpellier
  - UH NCaremeau, Nîmes